CLINICAL TRIAL: NCT02167412
Title: Electroencephalographic (EEG) Characteristics of Postural Tachycardia Syndrome (POTS) and Syncope (Without POTS) During Head-upright Tilt Table Testing
Brief Title: EEG Characteristics in Youth POTS and/or Syncope
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Heyer, MD, Nationwide Children's Hospital
Other Study IDs: IRB14-00252
Record Dates: First submitted 2014-06-13; First posted 2014-06-19 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Syncope; Postural Tachycardia Syndrome; Orthostatic Intolerance
Keywords: POTS; Syncope
MeSH Terms: conditions — Syncope; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Syncope without POTS: Patients meeting syncope criteria without POTS. There will be no intervention for this study arm.

SUMMARY:
Orthostatic intolerance refers to symptoms that occur with standing and improve or resolve with recumbency. Few studies have evaluated orthostatic intolerance symptoms by electroencephalography (EEG), and none of those studies have focused on the adolescent-aged patient. This study will compare EEG characteristics and sweat rate during head-upright tilt (HUT) testing among patients with postural tachycardia syndrome (POTS) and patients with syncope without POTS. Patients with POTS will also undergo a separate HUT with abdominal and lower extremity compression. The primary aim of this study is to characterize video EEG changes that correspond with orthostatic intolerance in youth during HUT testing. The investigators hypothesize that the clinical encephalopathy related to POTS and referred to as 'brain fog' will have an electrographic correlate. Secondary aims include (1) EEG comparisons of POTS symptoms with and without abdominal and lower extremity compression during HUT, (2) correlation between sweat rate and EEG changes during HUT, and (3) analysis of EEG characteristics that distinguish syncope with POTS from syncope without POTS. The investigators hypothesize that POTS patients have prolonged syncopal prodromes (compared to syncope patients without POTS) which are protective of syncope during daily activities.

DETAILED DESCRIPTION:
All POTS and syncope patients referred to Nationwide Children's Hospital (Columbus, OH) and meeting study eligibility criteria will be asked to participate. Consent and assent will be obtained per IRB guidelines. Consenting patients will undergo head-upright tilt (HUT) testing with video EEG and continuous sweat monitoring.

Prior to testing all medicines that can affect orthostatic tolerance will be held a minimum of 5 half-lives. Caffeine will be held for a minimum of 24 hours. Urinalysis (for urine specific gravity) and pregnancy testing (for female patients of child-bearing age) will be done the day of HUT testing. A recumbent EEG sample of no less than 10 minutes will be obtained. EKG leads, Holter leads, blood pressure monitors (beat-to-beat and conventional arm cuff), intravenous (IV) line, and sweat monitors will be placed. Sweat rate, EEG, and blood pressure monitoring will be synchronized by event trigger, allowing co-registration of all timed studies during data post-processing. Serum norepinephrine levels will be obtained at the time of IV placement and at 10 minutes of tilt or during/immediately after the syncope prodrome if syncope occurs prior to 10 minutes.

Once all monitors are placed, 10 minutes of EEG have been collected, and the patient has been recumbent for a minimum of 30 minutes, the table is tilted up-right to 70 degrees. A video camera will be on during the test. Patients are encouraged to report all symptoms and they are frequently examined for signs of pallor, acrocyanosis and sweating. Tilt testing is continued until syncope occurs, up to 10 minutes if the patient meets POTS criteria, or up to 45 minutes if neither syncope or POTS is not present.

Those who do meet age-appropriate POTS criteria (symptomatic heart-rate increment >40 bpm or symptomatic total HR of >130 bpm, all within 10 minutes of tilt for those <20 years of age) will be lowered at 10 minutes (or sooner with syncope) and asked to repeat testing with abdominal and lower extremity compression. The compression suit has been used by Dr. Heyer in other NCH studies. It is composed of a Neoprene-like material with 5 Velcro straps that fit snugly around the legs, thighs and abdomen. The abdominal strap contains an air-filled bladder that potentiates abdominal compression. We have used the suit in over 30 consenting patients from prior study. None of the study participants complained of discomfort. The suit successfully reduced both heart rate and orthostatic symptoms in youth with POTS; 55% of studied patients no longer met POTS diagnostic criteria while the suit was on (see PMID: 24840763 for manuscript). We will use the compression suit as our method of attenuating POTS symptoms during HUT testing. EEG will be compared without and with compression.

The time frame for this study is on average 90 minutes. It will not exceed 3 hours. After lowering the tilt table, all monitor leads and the IV will be removed. Once leads are removed there are no further study obligations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 9-21 years
* Referred to the neurology POTS and Syncope clinic at Nationwide Children's Hospital for clinical tilt table testing
* Has prior diagnosis or signs/symptoms of POTS (with or without syncope) or syncope (without POTS)

Exclusion Criteria:

* Cognitive, somatic or psychiatric illness that precludes tilt table testing, prolonged standing, or EEG lead placement
* Known seizure disorder
* Scalp or skull defect that could affect EEG amplitudes
* Pregnancy
* Non-English speaking

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred to the neurology-based POTS and Syncope clinic at Nationwide Children's Hospital (Columbus, OH) with POTS or with syncope without POTS and meeting eligibility criteria will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Video EEG characteristics of POTS and syncope | The time frame on average is 90 minutes and will not exceed 3 hours.
  Video EEG characteristics of orthostatic intolerance symptoms related to POTS (with and without syncope) and to syncope (without POTS) will be identified and compared between POTS and syncope cohorts.

SECONDARY OUTCOMES:
EEG characteristics of POTS with and without compression | The time frame on average is 90 minutes and will not exceed 3 hours.
  POTS patients will undergo two separate HUT tests, without and with abdominal and lower extremity compression. EEG characteristics will be compared between trials.
EEG comparison of syncopal prodrome with and without POTS | The time frame on average is 90 minutes and will not exceed 3 hours.
  EEG changes that correspond with the pre-syncopal prodrome (e.g., electrographic slowing) will be compared in terms of duration, quality of onset, and degree of change between syncope patients with and without POTS.
Correlation between sweat rate and EEG changes | The time frame on average is 90 minutes and will not exceed 3 hours.
  Orthostatic intolerance often has associated increases in sweat production. We will compare sweat rate and EEG changes in terms of temporal onset and peak changes to determine if sweat production correlates with EEG slowing.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L Heyer, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hopsital, Columbus, Ohio, United States

REFERENCES:
- See also: Nationwide Children's Hospital POTS and Syncope clinic — http://www.nationwidechildrens.org/postural-orthostatic-tachycardia-syndrome-clinic